CLINICAL TRIAL: NCT01903512
Title: Arthrocentesis and Temporomandibular Joint Disorders a Conservative Alternative to Surgical Treatments
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Silvio Mario Meloni, DDS, PhD, Assistant Professor, Università degli Studi di Sassari
Other Study IDs: IT010713
Record Dates: First submitted 2013-07-03; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: TMJ Internal Derangement
Keywords: TMJ arthrocentesis; internal derangement; conservative treatment
MeSH Terms: interventions — Arthrocentesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- arthrocentesis in TMJ internal derangement: 30 patients with TMJ internal derangement and pain with history of failed conservative management.
  Interventions: Procedure: TMJ arthrocentesis

INTERVENTIONS:
Procedure: TMJ arthrocentesis — lavage of the superior TMJ space with saline and sodium hyaluronate (SH)

SUMMARY:
This study aims to evaluate the efficacy of arthrocentesis in the treatment of internal derangement of the temporomandibular joint (TMJ).

DETAILED DESCRIPTION:
This work was designed as a prospective case series clinical study. Patients imaging was evaluated with Cone-Beam Computed Tomography and Nuclear Magnetic Resonance at the beginning of the treatment and after the last arthrocentesis.

ELIGIBILITY:
Inclusion Criteria:

* TMJ pain
* TMJ noises and click
* history of unsuccessful conservative management (NSAID and occlusal bite)
* occlusal bite still present

Exclusion Criteria:

* degenerative joint disease (such as osteoarthritis, rheumatoid arthritis etc.)
* history of condylar fractures or previous TMJ trauma
* TMJ surgery

Ages: 25 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 30 patients with TMJ internal derangement and pain with history of failed conservative management were selected. 70% had anteriorly displaced discs (AD), and 30 complained of other disorders (osteophytes, signs of soft tissues inflammmation, TMJ structure alterations).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pain decrease | baseline (preop), 1 week, 1 month, 2 months, 6 months, 12 months (postop)
  Patients were followed up for 1 year. The mean pre-operative pain, using visual analog scale, showed an average decrease of 6.7 at 1 year.
increase in the mouth opening | Baseline (preop), 1 week, 1 month, 2 months, 6 months, 12 months (postop)
  The mean maximum mouth opening(MMO) pre-operatively was 15,8 mm and increased to 34 mm immediately following arthrocentesis which increased by 0.5-1 mm at every month followup with mean MMO of 39,4 mm at 6 months. Thereafter it remained consistent till 1 year. The mean increase in the mouth opening at 1 year was 23,6 mm
TMJ click and noises reduction | Baseline (preop), 12 months (postop)
  At the end of 1 year, (75%) patients stated no evidence of clicking.

SECONDARY OUTCOMES:
number of subjects showing signs of TMJ inflammation or structural alterations at Magnetic Resonance Imaging and Cone Beam Computerized Tomography pre- and postop. | Baseline (preop)- 60 days postop
  40% of subjects who showed clear signs of inflammation showed significant improvement, in 30% with structural alterations was evident the absence of intra-articular adhesions and debris, in 30% with internal derangement did not appear any radiographic change.

CONTACTS AND LOCATIONS:
Overall Officials: Silvio M Meloni, assist prof, Principal Investigator — Università degli Studi di Sassari
Locations (1):
- Maxillofacial Unit, University of Sassari, Sassari, SS,, Italy

REFERENCES:
- [Derived] De Riu G, Stimolo M, Meloni SM, Soma D, Pisano M, Sembronio S, Tullio A. Arthrocentesis and temporomandibular joint disorders: clinical and radiological results of a prospective study. Int J Dent. 2013;2013:790648. doi: 10.1155/2013/790648. Epub 2013 Nov 11. PMID 24319462